CLINICAL TRIAL: NCT04273919
Title: A Pilot Study to Evaluate the Safety and Efficacy of the Karuna Virtual Reality Program for the Treatment of Chronic Low Back Pain
Brief Title: Virtual Reality for the Treatment of Chronic Low Back Pain
Acronym: VR
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the impact of COVID-19
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Michael Ashburn, MD, MPH, Director of Pain Medicine and Palliative Care, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 834277
Record Dates: First submitted 2020-02-04; First posted 2020-02-18 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Back Pain Lower Back Chronic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Mediation (Sham Comparator): Subjects will undergo virtual reality in a non-embodied (no first person bodily experience) program called Lumen, which was developed by Stanford University's Virtual Human Interaction Lab.
  Interventions: Device: HTC Vive with Lumen Program
- Graded Motor Imagery (Experimental): The subjects will engage in 2 therapeutic modules intended to help them practice increasing range of motion safely, and using small movements of the lower back.
  Interventions: Device: HTC Vive with Karuna Virtual Reality Program

INTERVENTIONS:
Device: HTC Vive with Karuna Virtual Reality Program — HTC Vive head-mounted display and an HTC Vive body tracker adhered to a belt on the patient's low back, which will be placed 2 inches below the waist
  Arms: Graded Motor Imagery
Device: HTC Vive with Lumen Program — HTC Vive head-mounted display with Lumen program
  Arms: Mindfulness Mediation

SUMMARY:
Chronic low back pain is highly prevalent in US adults and is a major cause of missed work days and disability. While several treatment options exist, chronic opioids are commonly used for these conditions even though there are limited data supporting efficacy, and clear evidence of harm associated with chronic opioid administration.

Virtual reality has been proposed as a treatment option that may lead to decreased pain and improved physical functioning, while avoiding the harms associated with medication management. This study is intended to obtain preliminary safety and efficacy data to guide the design of a larger clinical trial.

DETAILED DESCRIPTION:
This is a pilot study to evaluate the safety and efficacy of the Kauruna Virtual Reality program for the treatment of chronic low back pain. This study is intended to document the safety and efficacy of the use of virtual reality for the treatment of chronic low back pain. The primary outcome measure will be physical functioning as measured by the PROMIS 6. Secondary outcome measures include patient-reported pain intensity, adverse side effects, disability as measured by the Oswestry Low back disability questionnaire, and mental functioning as assessed using the PHQ-9 and GAD-7. Finally, impact on opioid use in patients on chronic opioids will be assessed by documentation of daily opioid dose in oral morphine equivalents.

Forty adult patients with chronic low back pain who are receiving care through the Penn Pain Medicine Center are eligible to participate in the study. The study will consist of a screening visit, followed by randomization into 1 of 2 study groups. Both study groups will participate in two 20-minute virtual reality sessions a week for 8 weeks. Study group 1 will participate in 20 minutes of mindfulness mediation. Study Group 2 will undergo initial sessions focused on graded motor imagery, followed by sessions focused on graded exposure. Patient-reported outcomes data will be obtained at baseline, then weekly during the 8-week study period, then 4 weeks following completion of the study sessions.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Able to speak and read English
* A history of chronic low back pain for at least 6 months
* No changes to medications within 30 days of randomization
* Able to provide outcomes data through the electronic patient-reported outcome data collection system

Exclusion Criteria:

* Age less than 18 years.
* Pregnant women
* Cognitive impairment that limits ability to participate in the study, including the provision of outcome data through the electronic patient-reported outcome data collection system.
* Unable to stand for at least 15 minutes
* Employees or students of the University of Pennsylvania

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Physical Functioning measured by PROMIS 6 (Patient Reported Outcome Measurement Information System) | 12 weeks
  Physical functioning reported on a scale 1 (unable to do) to 5 (without any difficulty)

SECONDARY OUTCOMES:
Patient-Reported Pain Intensity | 12 weeks
  Pain reported on a scale 0 (no pain) to 10 (worst pain possible)
Disability measured by the Oswestry Low Back Disability Questionnaire | 12 weeks
  Disability reported on a scale 0 (can complete task) to 5 (can't complete tasks)
Mental Functioning measured by PHQ-9 (Patient Health Questionnaire) | 12 weeks
  Mental functioning reported on a scale 0 (not at all) to 3 (nearly every day)
Mental Functioning measured by GAD-7 (Generalized Anxiety Disorder) | 12 weeks
  Mental functioning reported on a scale 0 (not at all) to 3 (nearly every day)
Adverse Events | 12 weeks
  Any symptom, sign, illness or experience that develops or worsens in severity during the course of the study will be documented

OTHER OUTCOMES:
Impact on opioid use | 12 weeks
  Impact on opioid use in patients on chronic opioids will be assessed by documentation of daily opioid dose in oral morphine equivalents.

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Ashburn, MD, MPH, Principal Investigator — Physician
Locations (1):
- Penn Pain Medicine Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Not applicable. Insufficient data collected. Study closed prematurely.

REFERENCES:
- See also: Karuna Labs FDA Establishment Registration — https://www.accessdata.fda.gov/scripts/cdrh/cfdocs/cfRL/rl.cfm?rid=211533